CLINICAL TRIAL: NCT01462045
Title: The Efficacy of Mindfulness-Based Stretching and Breathing Exercise as a Complementary Therapy for Posttraumatic Stress Disorder: A Prospective Randomized Study
Brief Title: Efficacy Study of Mindfulness-Based Exercise for Posttraumatic Stress Disorder (PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTSC027-2
Record Dates: First submitted 2011-10-07; First posted 2011-10-28 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2015-01-06 (Estimated); Status verified 2014-12

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: Exercise; Stress; PTSD; Mindfulness; Breathing; Cortisol
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity; Respiratory Aspiration | interventions — Breathing Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exercise Group (Experimental): Participants who are screened positive for PTSD and participate in the series of 16 standardized, semiweekly 60-minute mindfulness-based exercise sessions. The intervention consists of stretching and balancing movements combined with breathing and a focus on mindfulness.Over the course of 8 weeks, the intensity of the exercise increases, but the sequence of the movements is the same.
  Interventions: Behavioral: Mindfulness-based exercise
- Control Group (No Intervention): Participants who are screened positive for PTSD but do not participate in the mindfulness-based exercise.
- Base Group (No Intervention): Healthy volunteers who are not screened positive for PTSD and do not participate in the mindfulness-based exercise.

INTERVENTIONS:
Behavioral: Mindfulness-based exercise — 8-week program of mindfulness-based stretching and breathing exercises
  Other Names: Mindfulness stretching and breathing exercises
  Arms: Exercise Group

SUMMARY:
This study will explore the relationship between changes in plasma cortisol and symptom reduction resulting from individuals with posttraumatic stress disorder (PTSD) participating in an 8-week program of mindfulness-based stretching and breathing exercise. The investigators hypothesize that at the completion of participation in the 8-week program, exercise-induced symptom reduction will be associated with changes in cortisol levels.

DETAILED DESCRIPTION:
This study will employ an intent-to-treat design to evaluate the relationship between exercise-induced posttraumatic stress disorder (PTSD) symptom reduction and exercise-induced changes in cortisol level. The participants consist of nurses and the intervention will be conducted at the Clinical and Translational Science Center of the University of New Mexico. The study was approved by the Human Research Protections Office of the university. Nurses who are screened positively for PTSD will be randomly assigned to either control or exercise group. At baseline and in weeks 4, 8, 12 and 16, immediately after the phlebotomy for serum cortisol, the investigators will ask the participants to rate the severity of their PTSD symptoms using the PTSD Checklist (PCL).

ELIGIBILITY:
Inclusion Criteria:

* employed as a nurse
* PCL-C score of at least 28 with at least a score of 3 on one or more items for inclusion in the PTSD symptomatic groups (EX and CON)
* PCL-C score of 27 or lower for inclusion in the non-PTSD symptomatic group (BASE).

Exclusion Criteria:

* the inability to complete the exercise program
* a positive answer to any of the seven screening questions on the Physical Activity Readiness Questionnaire (PAR-Q)
* current use of prednisone or other forms of cortisone medication excluding cortisone in inhaled form

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Burge, MD, Principal Investigator — University of New Mexico
Locations (1):
- The University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Result] Kim SH, Schneider SM, Bevans M, Kravitz L, Mermier C, Qualls C, Burge MR. PTSD symptom reduction with mindfulness-based stretching and deep breathing exercise: randomized controlled clinical trial of efficacy. J Clin Endocrinol Metab. 2013 Jul;98(7):2984-92. doi: 10.1210/jc.2012-3742. Epub 2013 May 29. PMID 23720785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Nurse volunteers were recruited from the University of New Mexico Hospital through advertisement,between September 1, 2011 and March 31, 2012.
Pre-assignment Details: Participants gave their informed written consent before participation. Inclusion criteria were age greater than 18 years and employment as a nurse at the University of New Mexico (UNM) Hospital. Exclusion criteria included an inability to participate in the exercise program, or current use of systemic glucocorticoid.
Groups:
- Exercise Group: Participants who are screened positive for PTSD and participate in the mindfulness-based exercise.
Period: Overall Study
Arm/Group | Exercise Group | Control Group | Base Group
Started | 11 | 11 | 7
Completed | 11 | 10 | 7
Not Completed | 0 | 1 | 0
Not completed — Family matter | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise Group | Control Group | Base Group | Total
Number analyzed (Participants) | 11 | 11 | 7 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 6 | 28
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (6.4) | 45 (9.9) | 44 (15.1) | 46 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 7 | 28
  Male | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 7 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in PTSD Checklist - Civilian Version (PCL-C) Score
Description: The PCL-C is a 17-item self-report instrument that measures the symptoms of PTSD. A total score, ranging from 17 to 85, is found by summing the scores of the 17 items. Higher values are considered to be a worse outcome. The inclusion criteria in the PTSD symptomatic group is a PCL-C total score of at least 28 with a score of 3 or higher on 1 or more items.To detect a reduction in PTSD symptom severity with a 2-sided 5% significance level and a power of 80%, the mean difference of PCL-C scores of 5.16 or greater requires a sample size of 20 participants for Exercise and Control groups, given an anticipated dropout rate of 10%. Data analyses are conducted using an a priori intention-to-treat approach. The analysis for the between-group differences of the intervention is conducted using t-tests comparing Exercise and Control groups at post-intervention. The analysis for the within-group difference is conducted using repeated measures ANOVA for both groups at baseline and week 8.
Time Frame: Baseline and 8 weeks
Population: For Base Group, the values entered represent the mean value of the baseline PCL-C scores. The mean difference score for the Base Group is not available because the Base Group was assessed only at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Exercise Group | Control Group | Base Group
Number analyzed (Participants) | 11 | 11 | 7
scores on a scale | -18.8 (10.6) | -5.2 (15.8) | 21.8 (3.4)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = -13.6, 95% CI 2-sided [-25.6 to -1.6], Standard Error of Mean 5.7

2. Secondary Outcome: Cortisol
Description: Change from baseline in serum cortisol levels at 8 weeks. Serum cortisol samples were collected at 8:00 Ante Meridian (AM). The changes are calculated from two time points as the values at 8 weeks minus the values at baseline.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: μg/dl
Arm/Group | Exercise Group | Control Group | Base Group
Number analyzed (Participants) | 11 | 11 | 7
μg/dl | 5.1 (4.5) | -0.7 (6.5) | -0.04 (9.4)
Statistical Analysis 1: Comparison: Exercise Group vs Control Group; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; Mean Difference (Final Values) = 5.8, 95% CI 2-sided [0.83 to 10.8], Standard Error of Mean 2.4

ADVERSE EVENTS:
Arm/Group | Exercise Group | Control Group | Base Group
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No